CLINICAL TRIAL: NCT07389213
Title: Efficacy and Safety of rTMS Combined With HA in the Treatment of Cognitive Decline in Aged Related Hearing Loss: A Single-Center Real-World Study
Brief Title: Efficacy and Safety of rTMS Combined With HA in the Treatment of Cognitive Decline in Aged Related Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-525-01
Record Dates: First submitted 2025-11-25; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Senile Deadness
Keywords: senile deadness
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A total of 189 participants will be enrolled according to inclusion and exclusion criteria, including the ARHL-nonHA group, the ARHL-HA group, and the HC group. The three groups will undergo audiological assessments (PTA, SRT), cognitive function assessments (MoCA, MMSE, TMT-A, TMT-B, DST, SCWT), depression and sleep assessments (GDS-15, HAMD-24, PSQI), and imaging assessments (resting-state EEG, structural sMRI, resting-state functional rs-fMRI, task-based functional task-fMRI). The ARHL-nonHA and ARHL-HA groups will receive two courses of high-frequency rTMS stimulation, with each course lasting 14 days, one session per day, and each session lasting 9 minutes. Audiological, cognitive, depression and sleep, and imaging assessments will be performed on the ARHL-nonHA and ARHL-HA groups at 14 days and 1 month after the intervention, and the improvement values of the above indicators will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARHL-nonHA group (Experimental): This study will use repetitive transcranial magnetic stimulation (rTMS) as an intervention. Participants will be right-handed Chinese individuals aged between 50 and 85 years, diagnosed with moderate to severe age-related hearing loss (pure-tone average PTA of the better ear ranging from 35 to 79 dB), meeting the diagnostic criteria outlined in the 2019 expert consensus. Eligible participants must have at least 6 years of education and be able to complete all assessments in the Chinese version.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- ARHL-HA group (Experimental): This study will use repetitive transcranial magnetic stimulation (rTMS) as an intervention. Participants will be right-handed Chinese individuals aged between 50 and 85 years, diagnosed with moderate to severe age-related hearing loss (pure-tone average PTA of the better ear ranging from 35 to 79 dB).Participants must have been wearing hearing aids for more than six months and use them for over 7.2 hours daily. Eligible participants must have at least 6 years of education and be able to complete all assessments in the Chinese version.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- HC group (No Intervention): Aged between 50 and 85 years, with no gender restriction; pure-tone average (PTA) ≤25 dB HL in the better ear; Chinese nationality, able to complete all Chinese-version assessments; right-handed; and with at least 6 years of education.

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — High-frequency repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that modulates neural activity by delivering magnetic pulses to specific regions of the cerebral cortex. In this study, 50 Hz high-frequency stimulation will be used to enhance neuronal excitability, with stimulation intensity set at 80%-100% of the individual's motor threshold (MT) to accommodate the tolerance of elderly patients. Using each participant's MRI for neuronavigation, the stimulation coil will be precisely positioned over the left dorsolateral prefrontal cortex (DLPFC). Stimulation will be administered while the patient is awake, with each session lasting 9 minutes, delivered once daily. A single treatment course consists of 14 consecutive days, and a total of two courses will be conducted. Patient status will be closely monitored throughout the intervention to ensure safety and accuracy.
  Arms: ARHL-HA group; ARHL-nonHA group

SUMMARY:
This study is a real-world interventional trial enrolling 189 participants: older adults with age-related hearing loss not using hearing aids (ARHL-nonHA), those using hearing aids (ARHL-HA), and those with normal hearing (HC). All groups will undergo hearing, cognitive (MMSE, MoCA, SCWT, DST, TMT), depression (GDS-15, HAMD-24), sleep (PSQI), and brain imaging (EEG, sMRI, rs-fMRI, task-fMRI) assessments. The ARHL-nonHA and ARHL-HA groups will receive two 14-day courses of high-frequency rTMS (one session daily). One month after treatment, reassessments will be conducted in these two groups. Data will then be analyzed to evaluate the cognitive benefits of rTMS combined with hearing aids and to explore the underlying brain mechanisms.

DETAILED DESCRIPTION:
This study plans to conduct an interventional real-world study, enrolling 189 participants according to inclusion and exclusion criteria, including elderly patients with age-related hearing loss who do not wear hearing aids (ARHL-nonHA group), elderly patients with age-related hearing loss who wear hearing aids (ARHL-HA group), and elderly individuals with normal hearing (HC group). Audiological assessments (pure-tone average PTA, speech recognition threshold SRT), cognitive function assessments (Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Stroop Color-Word Test(SCWT), Digit Span Test (DST), Trail Making Test A (TMT-A), Trail Making Test B(TMT-B)), depression and sleep assessments (Geriatric Depression Scale (GDS-15), Hamilton Depression Rating Scale (HAMD-24), Pittsburgh Sleep Quality Index (PSQI)), and imaging assessments (resting-state (EEG), structural (sMRI), resting-state functional (rs-fMRI), task-based functional (task-fMRI)) will be performed on these three groups of participants. The ARHL-nonHA group and the ARHL-HA group will receive high-frequency repetitive Transcranial Magnetic Stimulation(rTMS) for two treatment courses, with each course lasting 14 days and one session per day. One month later, audiometric, cognitive, and imaging assessments will be repeated for the ARHL-nonHA and ARHL-HA groups. After the study, data will be collected and analyzed to evaluate the improvement effects of rTMS combined with HA on cognitive function in elderly patients with hearing loss, as well as its underlying brain functional mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years and ≤85 years, regardless of gender.
2. Diagnosed with age-related hearing loss (ARHL), characterized by symmetrical, slowly progressing hearing loss primarily affecting high frequencies, along with decreased speech recognition ability due to aging. This is in accordance with the "Expert Consensus on Diagnosis and Intervention of Age-Related Hearing Loss" 2019 edition.(Only ARHL-nonHA group and ARHL-HA group)
3. The better ear has moderate, moderately severe, or severe hearing loss (based on the 2021 WHO hearing classification standards, i.e., PTA between 35～79dB).
4. Wearing hearing aids for more than half a year, with daily wearing time exceeding 7.2 hours; (Only ARHL-HA group)
5. Chinese nationals who can complete all assessments in Chinese.
6. Right-handed.
7. Educational level of at least 6 years.
8. Informed consent obtained, agreeing to participate in the trial with no plans to relocate within one year.

Exclusion Criteria:

1. Exclusion of hearing loss due to noise, genetics, ototoxic drugs, or other non-age-related causes;
2. History of central nervous system disorders such as cerebral infarction, stroke, epilepsy, or traumatic brain injury;
3. Diagnosis of dementia or other neurodegenerative diseases that affect compliance with the study;
4. Presence of major neurological disorders, severe systemic diseases, family history of hereditary conditions, or major psychiatric disorders;
5. Contraindications to MRI;
6. Contraindications to rTMS.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment(MoCA ) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Montreal Cognitive Assessment (MoCA) ranges from 0 to 30, with higher scores indicating better cognitive function; a score of 26 or above is generally considered normal.
  The overall cognitive function in all groups with hearing loss was assessed using the MoCA scale before and after intervention, and the difference was calculated.

SECONDARY OUTCOMES:
Mini-Mental State Examination(MMSE) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Mini-Mental State Examination (MMSE) is scored on a scale from 0 to 30, with higher scores indicating better cognitive function.
  Overall cognitive function was assessed in all groups using the MMSE before and after the intervention, and the change scores were calculated.
Pure-Tone Average(PTA) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Pure-Tone Average (PTA) is calculated as the mean hearing threshold (in decibels hearing level, dB HL) at 500 Hz, 1 kHz, 2 kHz, and 4 kHz before and after intervention in the ARHL-HA group and the ARHL-nonHA group was assessed using pure-tone audiometry and sound field audiometry, and the difference was calculated.
Speech Reception Threshold(SRT) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Speech Reception Threshold (SRT) is the lowest intensity levelat which a person correctly identifies 50% of spondaic (two-syllable) words were correctly identified before and after intervention in the ARHL-HA group and the ARHL-nonHA group was assessed using speech audiometry and sound field speech audiometry, and the difference was calculated.
Trail Making Test Part A (TMT-A) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Trail Making Test Part A (TMT-A) is scored based on the time (in seconds) required to complete the task, with lower scores indicating better attention and information processing speed.
  The attention and information processing speed in the ARHL-HA group and the ARHL-nonHA group were assessed using the TMT-A before and after intervention, and the difference was calculated.
Trail Making Test Part B (TMT-B) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Trail Making Test Part B (TMT-B) is scored based on the time (in seconds) required to complete the task, with lower scores indicating better set-shifting ability and executive function.
  The set-shifting component of executive function in the ARHL-HA group and the ARHL-nonHA group was assessed using the TMT-B before and after intervention, and the difference was calculated.
Digit Span Test (DST)improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Digit Span Test (DST) is scored as the total number of correctly recalled digit sequences, with a typical total raw score ranging from 0 to 8. Higher scores indicate better attention, short-term memory, and working memory.
  Attention, short-term memory, and working memory in the ARHL-HA group and the ARHL-nonHA group were assessed using the DST before and after intervention, and the difference was calculated.
Stroop Color and Word Test (SCWT) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Stroop Color and Word Test (SCWT) is typically scored based on the time (in seconds) required to complete specific conditions .Lower completion times or lower interference scores indicate better inhibitory control and faster information processing speed, meaning lower values represent a better outcome.
  The inhibitory control of dominant responses and information processing speed, as components of executive function, in the ARHL-HA group and the ARHL-nonHA group were assessed using the SCWT before and after intervention, and the difference was calculated.
15-item Geriatric Depression Scale (GDS-15) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The 15-item Geriatric Depression Scale (GDS-15) is scored by summing the number of depressive symptom responses, with total scores ranging from 0 (no depressive symptoms) to 15 (most severe depressive symptoms). Higher scores indicate greater severity of depressive symptoms.
  Depressive symptom scores in the ARHL-HA group and the ARHL-nonHA group were assessed using the GDS-15 before and after intervention, and the difference was calculated.
24-item Hamilton Depression Rating Scale (HAMD-24)improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The 24-item Hamilton Depression Rating Scale (HAMD-24) is a clinician-administered measure of depressive symptom severity, with total scores ranging from 0 to 76. Higher scores indicate more severe depression.
  Depressive symptom scores in the ARHL-HA group and the ARHL-nonHA group were assessed using the HAMD-24 before and after intervention, and the difference was calculated.
Pittsburgh Sleep Quality Index (PSQI) improvement value | Baseline、Post-intervention 2 weeks and Post-intervention 1 month
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a one-month period. Total scores range from 0 to 21, with higher scores indicating poorer sleep quality.
  Sleep scores in the ARHL-HA group and the ARHL-nonHA group were assessed using the PSQI before and after intervention, and the difference was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Haidi, PhD, Study Chair — SunYatSunU2H
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China